CLINICAL TRIAL: NCT02207244
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo and Active Comparator-controlled Study Evaluating the Efficacy and Safety of Guselkumab for the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis With Randomized Withdrawal and Retreatment
Brief Title: A Study of Guselkumab in the Treatment of Participants With Moderate to Severe Plaque-Type Psoriasis With Randomized Withdrawal and Retreatment
Acronym: VOYAGE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR105048; CNTO1959PSO3002 (Other: Janssen Research & Development, LLC); 2014-000720-18 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-06

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque-type psoriasis; Guselkumab; Adalimumab; CNTO 1959; Monoclonal antibody
MeSH Terms: conditions — Psoriasis | interventions — guselkumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Participants will receive guselkumab 100 milligram (mg) at Weeks 0, 4, 12 and 20. Starting at Week 28, participants will receive guselkumab 100 mg or placebo through Week 72 depending upon randomized treatment group and PASI response. Placebo for guselkumab at Week 16, starting at Week 28, participants will continue to receive placebo for guselkumab through Week 72 depending upon randomized treatment group and PASI response. Placebo for adalimumab [two 0.8 milliliter (mL) injections] at Week 0 followed by one 0.8 mL injection at Weeks 1, 3, 5, and every 2 week (q2w) through Week 23 to maintain the blind. All participants will receive guselkumab q8w starting at Week 76 through Week 252.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Placebo for adalimumab
- Group II (Placebo Comparator): Participants will receive placebo for guselkumab at weeks 0, 4, 12 and starting at week 28 thereafter up to week 72 depending upon PASI response. Placebo for adalimumab (two 0.8 mL injections) at week 0, followed by one 0.8 mL injection at weeks 1, 3, and 5, and q2w through week 23. At week 16, placebo participants will cross over to receive guselkumab 100 mg at Weeks 16 and 20, starting at week 28, participants will continue to receive guselkumab 100 mg or placebo through week 72 depending upon PASI response. All participants will received guselkumab q8w starting at Week 76 through Week 252.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Placebo for adalimumab
- Group III (Active Comparator): Participants will receive adalimumab 80 mg (two 40 mg [0.8 mL] injections) at Week 0 followed by adalimumab 40 mg at weeks 1, 3, 5, and q2w through week 23 and placebo for guselkumab at weeks 0, 4, 12, 16, and 20. Participants will receive guselkumab or placebo starting at week 28 through week 72 depending upon PASI response. All participants will received guselkumab q8w starting at Week 76 through Week 252.
  Interventions: Drug: Guselkumab 100 mg; Drug: Placebo for guselkumab; Drug: Adalimumab

INTERVENTIONS:
Drug: Guselkumab 100 mg — 100 mg by subcutaneous injection at Weeks 0, 4, 12, and 20. Starting at Week 28, participants will continue to receive guselkumab 100 mg through Week 72 depending upon randomized treatment group and PASI response (Group I). 100 mg by subcutaneous injection at Weeks 16 and 20. Starting at Week 28, participants will continue to receive guselkumab 100 mg through Week 72 depending upon PASI response (Group II). Starting at Week 28, participants will receive guselkumab 100 mg through Week 72 depending upon PASI response (Group III). All participants will receive guselkumab q8w starting at Week 76 through Week 252.
  Other Names: CNTO 1959
Drug: Placebo for guselkumab — Placebo for guselkumab at Week 16, starting at Week 28, participants will continue to receive placebo for guselkumab through Week 72 depending on randomized treatment group and PASI response (Group I), at weeks 0, 4, 12 and starting at week 28 thereafter up to week 72 depending upon PASI response (Group II), at weeks 0, 4, 12, 16, and 20, starting at week 28 through week 72 depending upon PASI response (Group III).
Drug: Adalimumab — 80 mg by subcutaneous injection at Week 0, then 40 mg at Week 1 and every 2 weeks (q2w) thereafter through Week 23.
  Other Names: HUMIRA®
  Arms: Group III
Drug: Placebo for adalimumab — Placebo for adalimumab [two 0.8 milliliter (mL) injections] at week 0 followed by one 0.8 mL injection at weeks 1, 3, 5, and every 2 week (q2w) through Week 23 (Group I and II).
  Arms: Group I; Group II

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of guselkumab (CNTO 1959) in the treatment of participants with moderate to severe plaque-type psoriasis (scaly skin rash).

DETAILED DESCRIPTION:
This is a randomized (assignment of study drug by chance), double-blind (neither the participant or study staff will know the identity of study drugs), placebo- (inactive substance identical in appearance to study drug) and active-comparator-controlled (use of an approved drug to compare with study drug) study of guselkumab. The active comparator study drug is adalimumab, an approved drug for the treatment of moderate to severe plaque psoriasis. Participants who satisfy all inclusion and exclusion criteria will be randomly assigned in a 2:1:1 ratio to one of three treatment groups (arms): Group I (guselkumab 100 mg dose regimen), Group II (placebo then crossover to guselkumab at Week 16), or Group III (adalimumab at standard psoriasis dosing). From Week 28 up to Week 76, treatment for all participants will be based on their level of response. All participants will receive guselkumab every 8 weeks from Week 76 through Week 252 with a final safety follow-up visit at Week 264 (open label treatment period). The end of the study is defined as the time the last participant completes the Week 264 visit. The total duration of the study will be approximately 268 weeks (includes a 4-week screening period). Participants will be monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque-type psoriasis (with or without psoriatic arthritis) at least 6 months before the first administration of study agent
* Have a Psoriasis Area and Severity Index (PASI) greater than or equal to (>=) 12 at Screening and at Baseline
* Have an Investigator's Global Assessment (IGA) score >=3 at Screening and at Baseline
* Have an involved body surface area (BSA) >=10 percent (%) at Screening and at Baseline
* Must be a candidate for either systemic therapy or phototherapy for psoriasis

Exclusion Criteria:

* Participants with nonplaque forms of psoriasis (for example, erythrodermic, guttate, or pustular) or with current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* Participants who have ever received guselkumab or adalimumab
* History or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
* Is pregnant, nursing, or planning a pregnancy (both men and women) within 5 months following the last administration of study drug

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (93):
- United States (32):
  - Birmingham, Alabama
  - Bakersfield, California
  - Los Angeles, California
  - San Diego, California
  - Santa Monica, California
  - Aurora, Colorado
  - Coral Gables, Florida
  - Tampa, Florida
  - Newnan, Georgia
  - Sandy Springs, Georgia
  - Chicago, Illinois
  - Rolling Meadows, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Plainfield, Indiana
  - Louisville, Kentucky
  - Andover, Massachusetts
  - Fort Gratiot, Michigan
  - Troy, Michigan
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Gahanna, Ohio
  - Norman, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Johnston, Rhode Island
  - Arlington, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington
- Australia (6):
  - Benowa
  - Hectorville
  - Melbourne
  - Parkville
  - Westmead
  - Woolloongabba
- Canada (8):
  - Barrie, Ontario
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Richmond Hill, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
- Czechia (6):
  - Jihlava
  - Náchod
  - Pardubice
  - Pilsen
  - Prague
  - Ústí nad Labem
- Germany (9):
  - Dresden
  - Gera
  - Hamburg
  - Kiel
  - Leipzig
  - Lübeck
  - Münster
  - Tübingen
  - Witten
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lodz
  - Lublin
  - Olsztyn
  - Poznan
  - Torun
  - Warsaw
  - Wroclaw
- Russia (7):
  - Chelyabinsk
  - Cherepovets
  - Moscow
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Yaroslavl
- South Korea (7):
  - Busan
  - Daejeon
  - Gwangju
  - Incheon
  - Seongnam
  - Seoul
  - Suwon
- Spain (7):
  - Badalona
  - Barcelona
  - Bilbao Vizcaya
  - Madrid
  - Murcia
  - Pontevedra
  - Valencia

REFERENCES:
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Kim BS, Jo SJ, Youn S, Reich K, Saadoun C, Chang CL, Yang YW, Huang YH, Tsai TF. Five-year Maintenance of Clinical Response and Consistent Safety Profile for Guselkumab in Asian patients with Psoriasis from VOYAGE 1 and VOYAGE 2. Dermatol Ther (Heidelb). 2023 Nov;13(11):2721-2737. doi: 10.1007/s13555-023-01026-7. Epub 2023 Sep 26. PMID 37750995
- [Derived] Tillett W, Egeberg A, Sonkoly E, Gorecki P, Tjarnlund A, Buyze J, Wegner S, McGonagle D. Nail psoriasis dynamics during biologic treatment and withdrawal in patients with psoriasis who may be at high risk of developing psoriatic arthritis: a post hoc analysis of the VOYAGE 2 randomized trial. Arthritis Res Ther. 2023 Sep 15;25(1):169. doi: 10.1186/s13075-023-03138-z. PMID 37715294
- [Derived] Orbai AM, Chakravarty SD, You Y, Shawi M, Yang YW, Merola JF. Efficacy of Guselkumab in Treating Nails, Scalp, Hands, and Feet in Patients with Psoriasis and Self-reported Psoriatic Arthritis. Dermatol Ther (Heidelb). 2023 Nov;13(11):2859-2868. doi: 10.1007/s13555-023-01012-z. Epub 2023 Sep 15. PMID 37713133
- [Derived] Reich K, Gordon KB, Strober BE, Armstrong AW, Miller M, Shen YK, You Y, Han C, Yang YW, Foley P, Griffiths CEM. Five-year maintenance of clinical response and health-related quality of life improvements in patients with moderate-to-severe psoriasis treated with guselkumab: results from VOYAGE 1 and VOYAGE 2. Br J Dermatol. 2021 Dec;185(6):1146-1159. doi: 10.1111/bjd.20568. Epub 2021 Sep 8. PMID 34105767
- [Derived] Reich K, Armstrong AW, Foley P, Song M, Miller M, Shen YK, You Y, Han C, Gordon KB. Maintenance of Response Through up to 4 Years of Continuous Guselkumab Treatment of Psoriasis in the VOYAGE 2 Phase 3 Study. Am J Clin Dermatol. 2020 Dec;21(6):881-890. doi: 10.1007/s40257-020-00555-7. PMID 32910434
- [Derived] Gordon KB, Armstrong AW, Foley P, Song M, Shen YK, Li S, Munoz-Elias EJ, Branigan P, Liu X, Reich K. Guselkumab Efficacy after Withdrawal Is Associated with Suppression of Serum IL-23-Regulated IL-17 and IL-22 in Psoriasis: VOYAGE 2 Study. J Invest Dermatol. 2019 Dec;139(12):2437-2446.e1. doi: 10.1016/j.jid.2019.05.016. Epub 2019 Jun 15. PMID 31207232
- [Derived] Reich K, Papp KA, Armstrong AW, Wasfi Y, Li S, Shen YK, Randazzo B, Song M, Kimball AB. Safety of guselkumab in patients with moderate-to-severe psoriasis treated through 100 weeks: a pooled analysis from the randomized VOYAGE 1 and VOYAGE 2 studies. Br J Dermatol. 2019 May;180(5):1039-1049. doi: 10.1111/bjd.17454. PMID 30485400
- [Derived] Armstrong AW, Reich K, Foley P, Han C, Song M, Shen YK, You Y, Papp KA. Improvement in Patient-Reported Outcomes (Dermatology Life Quality Index and the Psoriasis Symptoms and Signs Diary) with Guselkumab in Moderate-to-Severe Plaque Psoriasis: Results from the Phase III VOYAGE 1 and VOYAGE 2 Studies. Am J Clin Dermatol. 2019 Feb;20(1):155-164. doi: 10.1007/s40257-018-0396-z. PMID 30417277
- [Derived] Foley P, Gordon K, Griffiths CEM, Wasfi Y, Randazzo B, Song M, Li S, Shen YK, Blauvelt A. Efficacy of Guselkumab Compared With Adalimumab and Placebo for Psoriasis in Specific Body Regions: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Dermatol. 2018 Jun 1;154(6):676-683. doi: 10.1001/jamadermatol.2018.0793. PMID 29799960

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Week 0 - 16): Participants received placebo matched to guselkumab subcutaneous (SC) injection at Weeks 0, 4, and 12 and placebo matched to adalimumab (2 SC injections) at Week 0, followed by placebo matched to adalimumab (1 SC injection) at Week 1 and every other week thereafter through Week 15 to maintain the blind during placebo controlled period (PCP).
- Guselkumab 100 mg (Week 0 - 16): Participants received guselkumab 100 milligram (mg) SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 followed by placebo matched to adalimumab (1 SC injection) at Week 1 and every other week thereafter through Week 15 during PCP.
- Adalimumab (Week 0 - 16): Participants received adalimumab 80 mg (2 SC injections) at Week 0 followed by adalimumab 40 mg (1 SC injection) at Week 1 and every other week thereafter through Week 15 and placebo matched to guselkumab SC injection at Weeks 0, 4, and 12 during PCP.
- Placebo Then Guselkumab 100 mg (Week 16 - 28): Participants who started receiving placebo in the first period were crossed over to receive guselkumab 100 mg SC injection at Weeks 16 and 20 and placebo matched to adalimumab (1 SC injection) at Weeks 17, 19, 21, and 23 during the active comparator controlled period (ACP).
- Guselkumab 100 mg (Week 16 - 28): Participants who started receiving guselkumab in the first period, received placebo matched to guselkumab SC injection at Week 16 followed by guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at Weeks 17, 19, 21 and 23.
- Adalimumab (Week 16 - 28): Participants who received adalimumab in the first period, continued to receive adalimumab 40 mg (1 SC injection) every 2 weeks (q2w) from Week 17 through Week 23 and placebo matched to guselkumab SC injection at Weeks 16 and 20.
- Placebo Then Guselkumab 100 mg (Week 28 - 264): Participants assigned to the placebo, then guselkumab arm through Week 28 were assessed for PASI 90 response at Week 28. Participants who were PASI 90 non-responders received guselkumab 100 mg SC injection at Week 28 and then every 8 weeks (q8w) thereafter through Week 72 and placebo matched to guselkumab SC injection at Week 32 and then q8w through Week 72. Participants who were PASI 90 responders at Week 28 received placebo matched to guselkumab SC injection at Week 28 and every 4 weeks (q4w) thereafter through Week 72 or until loss of greater than or equal to (>=) 50 percentage (%) in the improvement in PASI (Withdrawal and retreatment period). If they lost response according to this definition, they were retreated with guselkumab. Thereafter, participants received guselkumab 100 mg at Week 76 and then q8w through Week 252.
- Guselkumab 100 mg (Week 28 - 264): Participants assigned to the guselkumab arm through Week 28 were assessed for PASI 90 response at Week 28. Participants who were PASI 90 non-responders at Week 28 received guselkumab 100 mg SC injection at Week 28 and q8w thereafter through Week 72 and placebo matched to guselkumab at Week 32 and then q8w through Week 72. Participants who were PASI 90 responders were re-randomized to either guselkumab or placebo. Participants re-randomized to guselkumab, received guselkumab 100 mg SC injection at Week 28 and q8w thereafter through Week 72 and placebo matched to guselkumab SC injection at Weeks 32 and then q8w through Week 72. Participants re-randomized to placebo, received placebo matched to guselkumab SC injection q4w through Week 72 or until loss of >=50% in the improvement in PASI (Withdrawal and retreatment period). If they lost response according to this definition, they were retreated with guselkumab. Thereafter, participants received guselkumab 100 mg at Week 76 and then q8w through Week 252.
- Adalimumab Then Guselkumab 100 mg (Week 28 - 264): Participants who were assigned to the adalimumab arm through Week 28 were assessed for PASI 90 response at Week 28. Participants who were PASI 90 non-responders at Week 28 received guselkumab 100 mg SC injection at Week 28 and 32 and q8w thereafter through Week 72 and placebo matched to guselkumab SC injection at Weeks 36 and 44. Participants who were PASI 90 responders, received placebo matched to guselkumab SC injection q4w thereafter through Week 72 or until loss of >=50% in the improvement in PASI (Withdrawal and retreatment period). If they lost response according to this definition, they were treated with guselkumab. Thereafter, participants received guselkumab 100 mg at Week 76 and then q8w through Week 252.
- Adalimumab (After ACP): Participants who received adalimumab 80 mg at Week 0 and adalimumab 40 mg at Week 1 and every other week through Week 23 were assessed for PASI 90 response at Week 28. PASI 90 responders who did not crossover to guselkumab upon loss of >=50% in the improvement in PASI and did not continue any treatment at Week 28 are reported in this arm.
- Guselkumab Combined: All participants who received guselkumab 100 mg subcutaneously q8w at Week 76 and thereafter through Week 252.
Period: Placebo Controlled Period: Week 0-16
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 100 mg (Week 0 - 16) | Adalimumab (Week 0 - 16) | Placebo Then Guselkumab 100 mg (Week 16 - 28) | Guselkumab 100 mg (Week 16 - 28) | Adalimumab (Week 16 - 28) | Placebo Then Guselkumab 100 mg (Week 28 - 264) | Guselkumab 100 mg (Week 28 - 264) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) | Adalimumab (After ACP) | Guselkumab Combined
Started | 248 | 496 | 248 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 248 | 494 | 248 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 233 | 478 | 237 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 18 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 9 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — OTHER | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Placebo Crossover and ACP: Week 16-28
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 100 mg (Week 0 - 16) | Adalimumab (Week 0 - 16) | Placebo Then Guselkumab 100 mg (Week 16 - 28) | Guselkumab 100 mg (Week 16 - 28) | Adalimumab (Week 16 - 28) | Placebo Then Guselkumab 100 mg (Week 28 - 264) | Guselkumab 100 mg (Week 28 - 264) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) | Adalimumab (After ACP) | Guselkumab Combined
Started | 0 | 0 | 0 | 233 | 478 | 237 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 227 | 470 | 228 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 6 | 8 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Withdrawal and Re-treatment: Week 28-72
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 100 mg (Week 0 - 16) | Adalimumab (Week 0 - 16) | Placebo Then Guselkumab 100 mg (Week 16 - 28) | Guselkumab 100 mg (Week 16 - 28) | Adalimumab (Week 16 - 28) | Placebo Then Guselkumab 100 mg (Week 28 - 264) | Guselkumab 100 mg (Week 28 - 264) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) | Adalimumab (After ACP) | Guselkumab Combined
Started | 0 | 0 | 0 | 0 | 0 | 0 | 227 | 470 | 220 | 8 | 0
Nonresponders | 0 | 0 | 0 | 0 | 0 | 0 | 80 | 95 | 112 | 0 | 0
Responders at Week 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 375 (Participants randomized to withdrawal=182 and maintenance= 193) | 0 | 0 | 0
Responders at Week 28 and Withdrawn From Treatment (These participants were re-treated with guselkumab at or before Week 72.) | 0 | 0 | 0 | 0 | 0 | 0 | 147 | 0 | 108 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 213 | 443 | 211 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 27 | 9 | 8 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 3 | 2 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 2 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Participants not retreated with guselkumab | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Period: Open-label Guselkumab: Week 72-264
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 100 mg (Week 0 - 16) | Adalimumab (Week 0 - 16) | Placebo Then Guselkumab 100 mg (Week 16 - 28) | Guselkumab 100 mg (Week 16 - 28) | Adalimumab (Week 16 - 28) | Placebo Then Guselkumab 100 mg (Week 28 - 264) | Guselkumab 100 mg (Week 28 - 264) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) | Adalimumab (After ACP) | Guselkumab Combined
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 211 | 0 | 656
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 173 | 0 | 554
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 0 | 102
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 30
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 26
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 21
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 19
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo matched to guselkumab SC injection at Weeks 0, 4 and 12 and placebo matched to adalimumab (2 SC injections) at Week 0, followed by placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w thereafter through Week 15 to maintain the blind during PCP.
- Guselkumab 100 mg: Participants received guselkumab 100 mg SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5, and q2w thereafter through Week 15.
- Adalimumab: Participants received adalimumab 80 mg (2 SC injections) at Week 0 followed by adalimumab 40 mg (1 SC injection) at Weeks 1, 3, 5 and thereafter through week 15 and placebo matched to guselkumab SC injection at Weeks 0, 4, and 12.
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 100 mg | Adalimumab | Total
Number analyzed (Participants) | 248 | 496 | 248 | 992
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 3 | 0 | 8
  Between 18 and 65 years | 234 | 470 | 237 | 941
  >=65 years | 9 | 23 | 11 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.38) | 43.7 (12.23) | 43.2 (11.92) | 43.5 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 147 | 78 | 300
  Male | 173 | 349 | 170 | 692
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 13 | 25 | 13 | 51
  Czech Republic | 9 | 14 | 8 | 31
  Poland | 68 | 133 | 64 | 265
  Russia | 24 | 51 | 25 | 100
  Canada | 30 | 67 | 33 | 130
  United States | 49 | 93 | 48 | 190
  Germany | 22 | 40 | 22 | 84
  Spain | 10 | 22 | 11 | 43
  Korea, Democratic People'S Republic Of | 23 | 51 | 24 | 98

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Placebo Group at Week 16
Description: The IGA documents the investigator's assessment of the participants' psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 16
Population: Randomized analysis set included all participants who were randomized at Week 0. Nonresponder imputation (participants who met treatment-failure criteria before Week 16 or who did not come for evaluation at week 16 were considered nonresponders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Groups:
- Guselkumab 100 mg: Participants received guselkumab 100 mg SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w thereafter through Week 15.
Arm/Group | Placebo | Guselkumab 100 mg
Number analyzed (Participants) | 248 | 496
percentage of participants | 8.5 | 84.1
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

2. Primary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response in the Guselkumab Group Compared to the Placebo Group at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these area was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo matched to guselkumab SC injection at Weeks 0, 4 and 12 and placebo matched to adalimumab (2 SC injections) at Week 0, followed by placebo matched to adalimumab (1SC injection) at Weeks 1, 3, 5 and q2w thereafter through Week 15 to maintain the blind during PCP.
Arm/Group | Placebo | Guselkumab 100 mg
Number analyzed (Participants) | 248 | 496
percentage of participants | 2.4 | 70.0
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

3. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) in the Guselkumab Group Compared to the Adalimumab Group at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Randomized analysis set. Outcome measure was planned to be compared only for groups Guselkumab 100 mg and Adalimumab. Nonresponder imputation (participants who met treatment-failure criteria before Week 24 or who did not come for evaluation at Week 24 were considered nonresponders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Groups:
- Guselkumab 100 mg: Participants received guselkumab 100 mg SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w thereafter through Week 15. Participants received placebo matched to guselkumab SC injection at Week 16 then guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at Weeks 17, 19, 21 and 23.
- Adalimumab: Participants received adalimumab 80 mg (2 SC injections) at Week 0 followed by adalimumab 40 mg (1 SC injection) at Weeks 1, 3, 5 and every other week thereafter through Week 15 and placebo matched to guselkumab SC injection at Weeks 0, 4, and 12. Participants who received adalimumab in the first period, continued to receive adalimumab 40 mg (1 SC injection) q2w from Week 17 through Week 23 and placebo matched to guselkumab SC injection at Weeks 16 and 20.
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 51.8 | 31.5
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

4. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Adalimumab Group at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 83.5 | 64.9
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

5. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response in the Guselkumab Group Compared to the Adalimumab Group at Week 24
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 75.2 | 54.8
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

6. Secondary Outcome: Cumulative Maintenance Rate of Psoriasis Area and Severity Index (PASI) 90 Response in the Placebo Group Compared to the Guselkumab Group Through Week 48 to Evaluate Loss of a PASI 90 Response
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. Cumulative maintenance rate was defined as percentage of participants who maintained their PASI 90 response through Week 48.
Time Frame: Through Week 48
Population: Randomized analysis set included all participants who were randomized at Week 0 and who achieved a PASI 90 response at Week 28, were re-randomized to continue guselkumab or receive placebo and with at least one PASI assessment post Week 28.
Measure: Number; unit: Percentage of Participants
Groups:
- Withdrawal Group: Participants in withdrawal group received guselkumab 100 mg SC injection at Weeks 0, 4 and 12 and placebo matched to adalimumab (2 SC injections) at Week 0, followed by placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w through Week 15 to maintain the blind during PCP. Participants received placebo matched to guselkumab SC injection at Week 16 then guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at q2w from Week 17 through Week 23. These participants who were PASI 90 responders at Week 28 were randomized to receive placebo matched to guselkumab SC injection at Week 28 and q4w thereafter through Week 48 until loss of >=50% in the improvement in PASI.
- Guselkumab Maintenance Group: Participants of maintenance group received guselkumab 100 mg SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5, 7, and q2w through Week 15. Participants received placebo matched to guselkumab SC injection at Week 16 then guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at q2w from Week 17 through Week 23. These participants were PASI 90 responders who were randomized to receive guselkumab 100 mg SC injection at Week 28 and q8w thereafter through Week 44 and placebo matched to guselkumab SC injection at Weeks 32, 40 and 48.
Arm/Group | Withdrawal Group | Guselkumab Maintenance Group
Number analyzed (Participants) | 181 | 193
Percentage of Participants | 35.4 | 81.8
Statistical Analysis 1: Comparison: Withdrawal Group vs Guselkumab Maintenance Group; p value is based on the log-rank test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Log Rank

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Time Frame: Baseline, Week 16
Population: Randomized analysis set included all participants who were randomized at Week 0 and with a baseline DLQI score. Outcome measure was planned to be compared only for groups Placebo and Guselkumab 100 mg.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg
Number analyzed (Participants) | 248 | 495
units on a scale | -2.6 (6.85) | -11.23 (6.82)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; p value is based on analysis of variance (ANOVA) model stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, ANOVA

8. Secondary Outcome: Percentage of Participants Who Achieved an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab: Participants received adalimumab 80 mg (2 SC injections) at Week 0 followed by adalimumab 40 mg (1 SC injection) at Weeks 1, 3, 5 and every other week thereafter through Week 15 and placebo matched to guselkumab SC injection at Weeks 0, 4, and 12.
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 84.1 | 67.7
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on 1-sided Mantel Haenszel (MH) Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= -10.0%; p < 0.001, MH Z-test; Difference in Percentage = 16.4, 95% CI 2-sided [10.0 to 23.2]
Statistical Analysis 2: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

9. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response, in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: as for outcome 5
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 70.0 | 46.8
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on 1-sided MH Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= -10.0%; p < 0.001, MH Z-test; Difference in Percentage = 23.3, 95% CI 2-sided [16.0 to 30.4]
Statistical Analysis 2: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

10. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response in the Guselkumab Group Compared to the Adalimumab Group at Week 16
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score.
Time Frame: Week 16
Population: Randomized analysis set. Outcome measure was planned to be compared only for groups Guselkumab 100 mg and Adalimumab. Nonresponder imputation (participants who met treatment-failure criteria before Week 16 or who did not come for evaluation at week 16 were considered nonresponders) was used to impute missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 496 | 248
percentage of participants | 86.3 | 68.5
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on 1-sided MH Z-test adjusted for investigator site (pooled); Test type: Non-Inferiority or Equivalence — non-inferiority margin= -10%; p < 0.001, MH Z-test; Difference in percentage = 17.7, 95% CI 2-sided [11.4 to 24.4]
Statistical Analysis 2: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

11. Secondary Outcome: Percentage of Participants Who Achieved a Scalp-specific Investigator's Global Assessment (Ss-IGA) Score of 0 or 1 and at Least a 2-Grade Improvement From Baseline at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions were assessed in terms of the clinical signs of redness, thickness, and scaliness, which are scored on a 5-point scale ranging from 0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, and 4 = severe disease.
Time Frame: Week 16
Population: Population analyzed included only randomized participants who had an ss-IGA score greater than or equal to (>=) 2 at baseline. Outcome measure was planned to be compared only for groups Placebo and Guselkumab 100 mg.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg
Number analyzed (Participants) | 202 | 408
percentage of participants | 10.9 | 80.6
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

12. Secondary Outcome: Change From Baseline in Psoriasis Symptom and Sign Diary (PSSD) Symptom Score at Week 16 in the Guselkumab Group Compared to the Placebo Group
Description: The PSSD (24 hour version) is a patient-reported outcome (PRO) questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom [or Sign] score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease.
Time Frame: Baseline and Week 16
Population: PSSD analysis set included all those participants who had baseline PSSD scores as the average score of at least 4 days out of the 7 days prior to the Week 0 visit. Outcome measure was planned to be compared only for groups Placebo and Guselkumab 100 mg.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg
Number analyzed (Participants) | 198 | 411
units on a scale | -8.3 (23.67) | -40.4 (26.52)
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg; p value is based on ANOVA model stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, ANOVA

13. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Symptom and Sign Diary (PSSD) Symptom Score of 0 in the Guselkumab Group Compared to the Adalimumab Group at Week 24
Description: as for outcome 12
Time Frame: Week 24
Population: PSSD analysis set included all those participants who were randomized at Week 0 and had baseline PSSD score greater than 0. Outcome measure was planned to be compared only for groups Guselkumab 100 mg and Adalimumab.
Measure: Number; unit: Percentage of participants
Groups:
- Guselkumab 100 mg: Participants received guselkumab 100 mg SC injection at Weeks 0, 4 and1 2, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w thereafter through Week 15.
Arm/Group | Guselkumab 100 mg | Adalimumab
Number analyzed (Participants) | 410 | 200
Percentage of participants | 35.1 | 22.5
Statistical Analysis 1: Comparison: Guselkumab 100 mg vs Adalimumab; p value is based on the Cochran-Mantel-Haenszel chi-square test stratified by investigator site (pooled); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test

14. Secondary Outcome: Cumulative Maintenance Rate of PASI 90 Response in the Guselkumab Withdrawal Group Compared to the Guselkumab Maintenance Group Through Week 72 to Evaluate Loss of a PASI 90 Response
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. Cumulative maintenance rate was determined for participants who were withdrawn from study medication and who maintained guselkumab every 8 weeks dosing schedule and was defined as percentage of participants who maintained their PASI 90 response through Week 72.
Time Frame: Through Week 72
Population: Population analyzed included PASI 90 responders at Week 28 and who were randomized at Week 28 and treated with guselkumab. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Withdrawal Group: Participants in withdrawal group received guselkumab 100 mg SC injection at Weeks 0, 4 and 12 and placebo matched to adalimumab (2 SC injections) at Week 0, followed by placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5 and q2w through Week 15 to maintain the blind during PCP. Participants received placebo matched to guselkumab SC injection at Week 16 then guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at q2w from Week 17 through Week 23. These participants who were PASI 90 responders at Week 28 were randomized to receive placebo matched to guselkumab SC injection at Week 28 and q4w thereafter through Week 72 until loss of >=50% in the improvement in PASI.
- Guselkumab Maintenance Group: Participants of maintenance group received guselkumab 100 mg SC injection at Weeks 0, 4 and 12, and placebo matched to adalimumab (2 SC injections) at Week 0 then placebo matched to adalimumab (1 SC injection) at Weeks 1, 3, 5, 7, and q2w through Week 15. Participants received placebo matched to guselkumab SC injection at Week 16 then guselkumab 100 mg SC injection at Week 20 and placebo matched to adalimumab (1 SC injection) at q2w from Week 17 through Week 23. These participants were PASI 90 responders who were randomized to receive guselkumab 100 mg SC injection at Week 28 and q8w thereafter through Week 72 and placebo matched to guselkumab SC injection at Weeks 32, 40 and thereafter through Week 72.
Arm/Group | Withdrawal Group | Guselkumab Maintenance Group
Number analyzed (Participants) | 181 | 193
percentage of participants | 11.5 | 86

15. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Week 252
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Guselkumab Combined: All participants who crossed over to receive guselkumab 100 mg subcutaneously at Week 16 from placebo group and participants who were randomized to guselkumab 100 mg group at Week 0. Placebo crossover participants were included in the guselkumab column after crossover to guselkumab.
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 560 | 177
percentage of participants | 82.0 | 79.1

16. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Week 252
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 560 | 177
percentage of participants | 93.4 | 92.7

17. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of Cleared (0) or Minimal (1) at Week 252
Description: The IGA documents the investigator's assessment of the participants' psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participants' psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 559 | 177
percentage of participants | 85.0 | 83.1

18. Secondary Outcome: Percentage of Participants With a DLQI Score of 0 or 1 at Week 252
Description: The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. The DLQI was calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. Higher scores indicate more impact on quality of life of participants. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline DLQI score >1. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 550 | 173
percentage of participants | 71.1 | 69.9

19. Secondary Outcome: Percentage of Participants Who Achieved a PSSD Symptom Score of 0 at Week 252
Description: The PSSD (24-hour version) is a PRO questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Symptom score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline PSSD symptom score >0. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 460 | 145
percentage of participants | 42.0 | 36.6

20. Secondary Outcome: Percentage of Participants Who Achieved a PSSD Sign Score of 0 at Week 252
Description: The PSSD (24-hour version) is a PRO questionnaire designed and validated to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. It consisted of 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 (absent) to 10 (worst imaginable) numerical rating scales for severity. Items were averaged on the daily symptom score and sign score when at least 3 items (>=50 percentage of 5 items) on these scales are answered. The average value is converted into 0-100 scoring, such that Sign score = average value*10, where, 0= least severe and 100= most severe and higher score indicates more severe disease. As per planned analysis, participants from the baseline guselkumab group and the placebo crossover group were combined into a single guselkumab group for assessment of this outcome measure.
Time Frame: Week 252
Population: Population analyzed included participants who were randomized at Week 0 and treated with guselkumab with baseline PSSD sign score >0. The analysis was performed using observed data after applying treatment failure rules. Here, N (Number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab Combined | Adalimumab Then Guselkumab 100 mg (Week 28 - 264)
Number analyzed (Participants) | 461 | 145
percentage of participants | 31.0 | 24.1

ADVERSE EVENTS:
Time Frame: Baseline (Week 0) up to Week 264
Description: Safety analysis: all participants who were randomized at Week 0, received >=1 dose of study agent (partial or complete). Participants who discontinued treatment prematurely were followed for at least 12 weeks after last dose. Participants who discontinued in the previous period and had safety follow-up continuing in the current period, were counted in both the periods.
Groups:
- Adalimumab Then Guselkumab 100 mg (Week 28 - 264): Participants who were assigned to the adalimumab arm through Week 28 were assessed for PASI 90 response at Week 28. Participants who were PASI 90 non-responders received guselkumab 100 mg SC injection at Week 28 and 32 and q8w thereafter through Week 72 and placebo matched to guselkumab SC injection at Week 36 and q8w through Week 72. Participants who were PASI 90 responders, received placebo matched to guselkumab subcutaneous injection q4w thereafter through Week 72 or until loss of >=50% in the improvement in PASI. If they lost response according to this definition, they were treated with guselkumab. Thereafter, participants received guselkumab 100 mg at Week 76 and then q8w through Week 252. The presentation of data from the adalimumab group from Week 28 to Week 264 is divided into 2 arms (adalimumab then guselkumab 100 mg (Week 28 - 264) and adalimumab (After ACP) in order to represent exposure to 2 different active study agents (adalimumab vs guselkumab).
Arm/Group | Placebo (Week 0 - 16) | Guselkumab 100 mg (Week 0 - 16) | Adalimumab (Week 0 - 16) | Placebo Then Guselkumab 100 mg (Week 16 - 28) | Guselkumab 100 mg (Week 16 - 28) | Adalimumab (Week 16 - 28) | Placebo Then Guselkumab 100 mg (Week 28 - 264) | Guselkumab 100 mg (Week 28 - 264) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) | Adalimumab (After ACP)
Serious Adverse Events (participants affected / at risk) | 3/248 | 8/494 | 6/248 | 5/233 | 10/481 | 3/240 | 36/229 | 66/473 | 36/220 | 1/11
Other Adverse Events (participants affected / at risk) | 60/248 | 125/494 | 51/248 | 33/233 | 63/481 | 45/240 | 144/229 | 297/473 | 159/220 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=248) | Guselkumab 100 mg (Week 0 - 16) (N=494) | Adalimumab (Week 0 - 16) (N=248) | Placebo Then Guselkumab 100 mg (Week 16 - 28) (N=233) | Guselkumab 100 mg (Week 16 - 28) (N=481) | Adalimumab (Week 16 - 28) (N=240) | Placebo Then Guselkumab 100 mg (Week 28 - 264) (N=229) | Guselkumab 100 mg (Week 28 - 264) (N=473) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) (N=220) | Adalimumab (After ACP) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Submaxillary Gland Enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disseminated Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiv Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection Site Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pilonidal Cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0
Retroperitoneal Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vestibular Neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nerve Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal Cord Injury Cervical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ulnar Nerve Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inflammatory Pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinonasal Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebellar Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelitis Transverse (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral Nerve Lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral Nerve Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device Dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Miscarriage of Partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0 - 16) (N=248) | Guselkumab 100 mg (Week 0 - 16) (N=494) | Adalimumab (Week 0 - 16) (N=248) | Placebo Then Guselkumab 100 mg (Week 16 - 28) (N=233) | Guselkumab 100 mg (Week 16 - 28) (N=481) | Adalimumab (Week 16 - 28) (N=240) | Placebo Then Guselkumab 100 mg (Week 28 - 264) (N=229) | Guselkumab 100 mg (Week 28 - 264) (N=473) | Adalimumab Then Guselkumab 100 mg (Week 28 - 264) (N=220) | Adalimumab (After ACP) (N=11)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 11 | 4 | 0 | 3 | 3 | 11 | 15 | 12 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 12 | 4 | 1
Bronchitis (Infections and infestations) | 3 | 3 | 5 | 6 | 3 | 3 | 15 | 23 | 21 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 5 | 0 | 1 | 0 | 11 | 16 | 11 | 0
Nasopharyngitis (Infections and infestations) | 16 | 35 | 20 | 12 | 18 | 16 | 67 | 142 | 81 | 0
Pharyngitis (Infections and infestations) | 2 | 7 | 1 | 2 | 5 | 2 | 18 | 32 | 5 | 0
Sinusitis (Infections and infestations) | 3 | 3 | 2 | 1 | 3 | 2 | 16 | 23 | 11 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 16 | 4 | 5 | 12 | 6 | 39 | 111 | 49 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 6 | 0 | 1 | 0 | 1 | 7 | 19 | 12 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 4 | 9 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 11 | 2 | 0 | 8 | 6 | 17 | 46 | 22 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0 | 6 | 0 | 18 | 25 | 16 | 1
Headache (Nervous system disorders) | 7 | 25 | 5 | 5 | 6 | 4 | 9 | 31 | 17 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 1 | 1 | 2 | 2 | 10 | 16 | 13 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 0 | 2 | 0 | 2 | 11 | 6 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 5 | 0 | 1 | 1 | 3 | 8 | 9 | 1
Hypertension (Vascular disorders) | 4 | 10 | 6 | 1 | 4 | 1 | 27 | 43 | 20 | 0

LIMITATIONS AND CAVEATS:
All participants were on guselkumab after Week 76; therefore, there was no concurrent control group within the study after Week 76.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.